CLINICAL TRIAL: NCT06103136
Title: Maestro 1.1 Post-Market Registry
Status: Recruiting | Type: Observational
Sponsor: Moon Surgical (Industry)
Responsible Party: Sponsor
Other Study IDs: Maestro1.1 PostMarket Registry
Record Dates: First submitted 2023-10-17; First posted 2023-10-26 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Surgery
Keywords: abdominal laparoscopic surgery; surgical assistance device

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Patients operated using the Maestro platform
  Interventions: Device: Laparoscopic surgery using the Maestro Platform
- Control
  Interventions: Device: Laparoscopic surgery using the Maestro Platform

INTERVENTIONS:
Device: Laparoscopic surgery using the Maestro Platform — Patients scheduled for laparoscopic surgery will be operated on as per standard of care, using standard port, surgical table and instrument placements (following local applicable guidelines), and off-the-shelf surgical equipment. Standard of care surgical technique following local applicable guidelines will be used.
  The Maestro Platform may be used to position and hold the scope as well as the retractor in the locations determined by the surgeon during the procedure, with the ability to revert at any time to standard of care (manual minimally invasive surgery) without the usage of the Maestro Platform, or to convert to open surgery.

SUMMARY:
The objective of the study is to observe the real-life usage of the Maestro Platform for surgical assistance in laparoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be adults aged ≥ 18 years scheduled for laparoscopic surgery.

Exclusion Criteria:

* Participants might be excluded based on the investigator's discretion.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General population scheduled for laparoscopic surgery.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-09-29 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AEs) in terms of type (device/procedure related), seriousness, level of severity. Rate of occurence of intra-procedural and post-procedural adverse events, and device related complications | Adverse Events (AEs) in terms of type (device/procedure related), seriousness, level of severity. Rate of occurence of intra-procedural and post-procedural adverse events, and device related complications [ Time Frame: 30 days ]
Completion of the procedure using the Maestro Platform without conversion to a manual minimally invasive or open surgical procedure specifically due to a device failure or malfunction | During procedure

SECONDARY OUTCOMES:
Incidence of procedure-specific complications | During procedure
Procedure duration | During procedure
Wheels-in Wheels-out | During procedure
  Timing and durations of Maestro's use in the procedure
Skin to Skin time | During procedure
  Duration between the first incision and the last suture
Recovery time | 30 days
  Assess whether the patient has fully recovered after 30 days
Turnaround time | During Procedure
  Time between the start of two interventions compared to a baseline without the use of the Maestro System
Camera cleaning rate | During procedure
  the rate at which the surgeon extracts the endoscope from the patient to clean it
Post operative pain | 1 day after the procedure
  Visual analogue scale 0 - no pain to 10 - worst pain possible
Potential post-operative complications | 30 days
Human resource utilization for surgical assistance in the operating room | During procedure
  Number and type of staff in the OR during the procedure
Surgeon comfort evaluated on 1-5 scale at the end of the procedure | During procedure
  1 - not comfortable 5 - very comfortable
Surgeon satisfaction with Maestro evaluated on 1-5 scale at the end of the procedure | During procedure
  1 - not satisfied 5 - very satisfied
Registry device preparation duration | During procedure

CONTACTS AND LOCATIONS:
Locations (12):
- United States (6):
  - Rose Medical Center, Denver, Colorado
  - Lee Health, Fort Myers, Florida
  - Baptist Health, Jacksonville, Florida
  - Baptist Medical Center Beaches, Jacksonville, Florida
  - Orlando Veterans Affairs Medical Center, Orlando, Florida
  - Surgeon's Point ASC, Cedar Park, Texas
- Chirec Delta, Auderghem, Belgium
- France (5):
  - Hôpital Privé Arnault Tzanck, Mougin, Alpes Maritimes
  - Polyclinique de Franche-Comté, Besançon
  - Clinique Bouchard, Marseille
  - Institut Arnault Tzanck, Saint-Laurent-du-Var
  - Clinique de l'Orangerie, Strasbourg

IPD SHARING:
Plan to Share IPD: Undecided